CLINICAL TRIAL: NCT02324075
Title: Using Behaviour Change Messaging to Improve Communal Toilets in Dhaka, Bangladesh
Acronym: WSUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Stephen P Luby, Primary Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPO-113016
Record Dates: First submitted 2014-11-11; First posted 2014-12-24 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Diarrhea
Keywords: sanitation, toilet, urban, behavior change
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavior change (Experimental): Behavior change messaging with facilitating hardware
  Interventions: Behavioral: Behavior change
- Control Arm (No Intervention): Standard habits and practices

INTERVENTIONS:
Behavioral: Behavior change — Non governmental organization delivers communication intervention with facilitating hardware, a waste bin and bucket
  Arms: Behavior change

SUMMARY:
Background (brief):

1. Burden: In low income neighborhoods in Dhaka many households share toilets which are often unsanitary and their discharge contaminates the community.
2. Knowledge gap: Behavior change messages have the potential to make people concerned about maintaining shared toilets quality, cleanliness and safety of the facility. There are many contributors to poor sanitation in low income neighborhoods in Dhaka but it's not clear that the situation can be improved with behavior change or even which specific messages to target.
3. Relevance: Water Sanitation for the Urban Poor (WSUP) is a nongovernmental organization working to improve shared sanitation facilities in Dhaka. They are interested in developing and evaluating a behavior change program to improve shared sanitation in Dhaka and to generate lessons that would be relevant for other low income urban settings globally.

Hypothesis: A behavior change communication intervention can improve the quality and cleanliness of sanitation services available to low-income residents of Dhaka.

Objectives:

1. To deliver behavior change messages (which target key behaviors influencing the quality and cleanliness of shared sanitation facilities) to randomly selected low-income communities in Dhaka.
2. To evaluate the effectiveness of a behavior change communication intervention designed to change targeted behaviors related to the quality and cleanliness of shared sanitation facilities.

Methods:

Local non-governmental organizations will deliver the intervention (behavior change communication package) in randomly selected communities. For this study the investigators will assess the impact of this intervention on the targeted behaviors using follow-up surveys and spot checks.

DETAILED DESCRIPTION:
Hypothesis to be tested: A behavior change communication intervention can improve the quality and cleanliness of sanitation services available to low-income residents of Dhaka.

Specific Objectives:

1. To deliver communication messages (selected as the most promising for changing target behaviors influencing the quality and cleanliness of shared sanitation facilities) to randomly selected low-income communities in Dhaka.
2. To evaluate the effectiveness of a behavior change communication intervention designed to change targeted behaviors related to the quality and cleanliness of shared sanitation facilities.

Background The investigators contend that important barriers to improved sanitation in low-income communities in Dhaka include: 1) Low-income community residents lack the financial resources to purchase a better option. 2) The cost of land in Dhaka, which has increased 600 fold since the 1970s (Hossain, 2011), makes space for toilets expensive 3) A public sector characterized by weak institutions that lack funding and management capacity to implement and maintain effective sanitary infrastructure (Hossain, 2011) and 4) a pervasive informal local political system that maximizes the financial interests of politically connected elites over the communal interests of low-income community residents (Hackenbroch and Hossain, 2012, Hossain, 2011). More than one third of Dhaka residents live in informal settlements where government authorities do not accept responsibility for providing urban utilities including water and sanitation services (World Bank, 2007). A central motivation for politicians to avoid formalizing settlements is that informality keeps residents in a constant state of dependency on local party associates, a state which these local elites can use to extract a continuous stream of resources (Anjaria, 2006, Hossain, 2011).

Behavior change communication messages cannot directly resolve these major barriers to improving community sanitation in low-income communities in Dhaka. Simple general messages, such as encouraging people to clean keep their sanitary facility clean to reduce the risk of disease transmission, are unlikely to be effective because they do not address the determinants of the poor availability, cleanliness and maintenance of shared sanitary facilities. By contrast, by developing behavior change messages that are informed by the experience and perspective of the target population this study can identify some opportunities where new information or a new social norm could alter some key behaviors.

The pilot work found considerable interest in cleaner better maintained latrines. Inclusion of 2 low-cost hardware accessories, a waste bin so that materials such as condoms or sanitary pads can be discarded in ways that do not block the toilet and bucket to assist with rinsing the toilet after defecation makes it easier for communities to follow behavior change recommendations to support a cleaner shared latrine.The central question for this research project is: Can a strategically designed behavior change campaign supplemented with low-cost hardware accessories shift the current equilibrium of unhygienic shared sanitation facilities towards cleaner facilities in low-income communities of Dhaka?

Research Design and Methods:

SUMMARY:

* Deliver behavior change communication messages using a behavior change communication intervention to randomly selected low-income communities in Dhaka. (Package of behavior change interventions for targeted behaviors: waste disposal, rules for latrine use and repair and maintenance)
* Evaluate the effectiveness of the behavior change communication intervention in changing the targeted behaviors.

DETAILS:

o Deliver messages using a behavior change communication intervention to randomly selected low-income communities in Dhaka.

The study team will add intervention components onto existing NGO interventions to increase impact and decrease cost. Thus, through extensive piloting informative work, the investigators have developed behavior change communication materials, based on specific behaviors targeted to improve latrine cleanliness and quality. The materials and messages will be used to train community health promoters (CHPs) that are currently working for the selected NGOs. Some materials will include sign boards for latrines that will be fixed to those areas randomly selected to receive the intervention. The intervention will also include enabling hardware, a waste bin for trash collection and the bucket for carrying water to flush the latrine. The intervention: these will be delivered by partner NGO community hygiene promoters. This intervention approach is aimed to leverage existing intervention delivery partners and thus add value across the sector. The investigators have identified an NGO partner with large urban programs including sanitation activities in Mirpur, Mohakhali and Mohammadpur.

The survey team will work with partner NGOs and identify the coverage areas that are eligible for participation in the study. These include:

1. Some larger slums with 60 to 180 communal toilets and sanitation interventions provided by 3 to 12 community health promoters whose activities collectively cover the entire slum area.
2. Some smaller slums with 6-10 communal toilets available for around 150 to 300 households. These communal toilets were situated very close to one another, and this type of slum is served by a single community health promoter.
3. Some scattered slums which are very small compared to other slums. This type of slum consists of 15-50 households sharing one communal toilet. One community health promoter covers 4-8 scattered slums.

The team will divide those selected slums into distinct clusters primarily based on community health promoter coverage area. If the area is very large, the CHP coverage areas will be sub-divided using geographic boundaries such as roads, bazaars, water bodies that clearly distinguish between distinct clusters. Each cluster will comprise:

1. an area covered by a single CHP
2. between 1 and 30 communal toilets

A communal toilet consists of a structure with approximately 2 to 16 chambers that drain into a common septic tank. The clusters will be the unit of randomization for this study.

At the beginning of the study, the study team will conduct a communal toilet listing to collect information on numbers of toilet users for each communal toilet. Once listing is done, a statistician who is independent of this project will randomly assign clusters to either the intervention or comparison arms. Clusters are separated geographically by streets, bazaars, fields, drainage or other settlements, and therefore investigators do not expect intervention messages or activities to spill over into control toilet clusters even when they are located very close by.

For each intervention cluster, the field will also enroll a matched control cluster, matched on the number of toilet chambers per cluster. Investigators will use the following categories for matching: <5 chambers, 5-10 chambers, 11-15 chambers, 16-20 chambers, and >20 chambers assuming that based on the number of chambers, the numbers of users could vary. A statistician, who is not a resident of Bangladesh and who is not a member of the study project, will randomly assign clusters to intervention versus control. WSUP, on behalf of the intervention team, will sign contracts with the partner NGOs to implement the behavior change package. The behavior change messages and enabling hardware will be delivered by the partner NGOs through their community health promoters (CHPs). Investigators will help partner NGOs train CHPs in the components of the intervention to ensure that CHPs conduct group meetings and inter-personal communication that will effectively convey our intervention messages.

The partner NGO will receive final behavior change communication materials from the study team and it will be responsible for printing and distribute these materials only to intervention communities. The research team will be involved with the implementation team to ensure that rollout occurs in the specified intervention clusters at the planned frequency and timing and that there is no messaging in the control clusters. Investigators will explain the plan for the fidelity assessment with the implementers and share the results as soon as they are available.

• Evaluate the effectiveness of the behavior change communication intervention in changing the targeted behaviors.

Behavior change campaigns that provoke discussion between viewers of the campaign and their social network are more likely to result in behavior change (Boulay et al., 2002, Hafstad and Aaro, 1997). The survey instrument includes objective uptake indicators, a measurement of exposure to the intervention, awareness of the behavior change package, frequency of discussion of the contents of the behavior change communication information with the respondent's social network, access to sanitation facilities and attitudes regarding the acceptability and cleanliness of these facilities. Investigators will conduct a pre-intervention baseline survey by drawing a systematic random sample of one adult user per communal toilet in both intervention and control clusters. The field team will sample equal numbers of users from intervention and control arms. The field team will visit the communal toilet and enroll the third household nearest to that communal toilet and administer the toilet user survey to one adult resident. If the selected user doesn't want to participate in the survey, the field team will approach a subsequent household for enrollment and also record the non-response. The field team will administer a toilet quality/cleanliness observation instrument to assess the primary objective indicators for all study toilets. To ensure inter-rater reliability of toilet observations among observers, a subset of communal toilet will be evaluated by two separate observers. Observer pairs will conduct their assessments during a 5-10 minutes interval, and their independent evaluations will be compared to make sure that our observers measure cleanliness consistently and objectively. Such research reliability observations will be conducted for initial 50 communal toilets, or until observer credibility can be effectively established and discrepancies minimized.

Along with quantitative survey, field investigators will also explore local elite or landlord's view on their role and roles of others in constructing, maintaining, cleaning and emptying the communal toilet facilities by conducting qualitative interviews for the previously mentioned three types of slums. Field investigators will conduct in-depth interview with 4 different landlord or elite from mentioned each types of slums or they will interview until they have reached data saturation. Field investigators will interview those elites or landlords before the intervention commences and at the end of the intervention.

The study team will conduct a baseline evaluation in intervention and control communities as well as an endline after the 6 months of intervention roll out. In addition, two months after initiation of the intervention, the field team will conduct a rapid fidelity assessment using the same survey instrument in a random subset of 50 intervention toilets. The purpose of this rapid assessment is to ensure that the behavior change intervention exposure is occurring at the expected level. If not, then the partner NGOs will be contacted and the problems addressed.

The study team will compare the change in targeted behaviors observed in the intervention communities compared with changes observed in the control communities and so measure the amount of behavior change attributable to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Residents of low income communities in Dhaka who share toilet facilities with non-family members

Exclusion Criteria:

* Special groups whose ability to give voluntary informed consent might be compromised

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1226 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: STEPHEN P LUBY, M.D., Principal Investigator — Stanford University
Locations (1):
- Icddr,B, Dhaka, Bangladesh

REFERENCES:
- [Result] Alam MU, Winch PJ, Saxton RE, Nizame FA, Yeasmin F, Norman G, Masud AA, Begum F, Rahman M, Hossain K, Layden A, Unicomb L, Luby SP. Behaviour change intervention to improve shared toilet maintenance and cleanliness in urban slums of Dhaka: a cluster-randomised controlled trial. Trop Med Int Health. 2017 Aug;22(8):1000-1011. doi: 10.1111/tmi.12902. Epub 2017 Jun 29. PMID 28556458
- [Result] Saxton RE, Yeasmin F, Alam MU, Al-Masud A, Dutta NC, Yeasmin D, Luby SP, Unicomb L, Winch PJ. If I do not have enough water, then how could I bring additional water for toilet cleaning?! Addressing water scarcity to promote hygienic use of shared toilets in Dhaka, Bangladesh. Trop Med Int Health. 2017 Sep;22(9):1099-1111. doi: 10.1111/tmi.12914. Epub 2017 Jul 25. PMID 28656596
- [Result] Yeasmin F, Luby SP, Saxton RE, Nizame FA, Alam MU, Dutta NC, Masud AA, Yeasmin D, Layden A, Rahman H, Abbott R, Unicomb L, Winch PJ. Piloting a low-cost hardware intervention to reduce improper disposal of solid waste in communal toilets in low-income settlements in Dhaka, Bangladesh. BMC Public Health. 2017 Aug 29;17(1):682. doi: 10.1186/s12889-017-4693-x. PMID 28851334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this cluster trial, communities were randomized either to receive a behavior change messaging intervention or no intervention. 1226 shared latrines were analyzed within these communities. One person using the shared latrine was asked to complete study surveys (baseline and month 6), and respondents were considered to be enrolled in the study.
Units Other Than Participants: Shared latrines
Period: Overall Study
Arm/Group | Behavior Change | Control Arm
Started | 612; 612 Shared latrines | 614; 614 Shared latrines
Completed | 609; 605 Shared latrines | 605; 605 Shared latrines
Not Completed | 3; 7 Shared latrines | 9; 9 Shared latrines

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavior Change | Control Arm | Total
Number analyzed (Participants) | 612 | 614 | 1226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 612 | 614 | 1226
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (11) | 34 (13) | 33.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 452 | 461 | 913
  Male | 160 | 153 | 313
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Bangladesh | 612 | 614 | 1226

OUTCOME MEASURES:

1. Primary Outcome: Number of Pans With Presence of Visible Feces Inside the Pan
Description: Assessment by observer in unannounced visit to the shared latrine to determine presence of visible feces inside the pan (both inside and outside the hole in the pan).
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle with waste pan. Pans that were evaluated were included in the analysis.
Measure: Count of Units; unit: pans
Units Other Than Participants: pans
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (pans) | 912 | 883
pans
  Baseline: number analyzed (pans) | 907 | 876
  Baseline | 282 | 203
  Month 6 | 83 | 124

2. Secondary Outcome: Number of Pans With Presence of Visible Feces Outside the Pan
Description: Assessment by observer in unannounced visit to the shared latrine to determine presence of visible feces outside the pan.
Time Frame: Assessed at 6 months post intervention
Population: as for outcome 1
Measure: Count of Units; unit: pans
Units Other Than Participants: pans
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (pans) | 912 | 883
pans
  Baseline: number analyzed (pans) | 907 | 876
  Baseline | 68 | 64
  Month 6 | 21 | 31

3. Secondary Outcome: Visible Feces on the Path Leading up to the Latrine
Description: Assessment by observer in unannounced visit to the shared latrine to determine presence of feces on the path leading up to the shared toilet.
Time Frame: Assessed at 6 months post intervention
Measure: Count of Units; unit: Shares latrines
Units Other Than Participants: Shares latrines
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Shares latrines) | 612 | 614
Shares latrines
  Baseline | 57 | 72
  Month 6 | 55 | 56

4. Secondary Outcome: Visible Feces Near the Latrine But Not on the Path
Description: Assessment by observer in unannounced visit to the shared latrine to determine presence of feces near the latrine but not on the path leading to the latrine.
Time Frame: baseline and 6 months post intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Functional Cubicle Toilets
Description: Assessment by observer in unannounced visit to the shared latrine to determine if the cubicle toilet is fully functional.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle toilet. Toilets that were evaluated were included in the analysis.
Measure: Count of Units; unit: toilets
Units Other Than Participants: toilets
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (toilets) | 919 | 935
toilets
  Baseline | 906 | 916
  Month 6: number analyzed (toilets) | 892 | 909
  Month 6 | 877 | 877

6. Secondary Outcome: Visible Feces Inside the Hole of the Pan
Description: Observer in unannounced visit assess if feces is visible inside the hole of the pan
Time Frame: Assessed at 6 months post intervention
Population: as for outcome 1
Measure: Count of Units; unit: pans
Units Other Than Participants: pans
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (pans) | 912 | 883
pans
  Baseline: number analyzed (pans) | 907 | 876
  Baseline | 433 | 399
  Month 6 | 297 | 351

7. Secondary Outcome: Latrine Cleanliness - Spit/Cough on Walls/Doors
Description: Assessment by observer in unannounced visit to the shared latrine to determine problems with cleanliness. Observations were made for spit/cough on walls/doors. The count of units that had the problem is presented for each problem type.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle. Cubicles that were evaluated were included in the analysis.
Measure: Count of Units; unit: Cubicles
Units Other Than Participants: Cubicles
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Cubicles) | 908 | 876
Cubicles
  Spit/cough on walls/doors (baseline): number analyzed (Cubicles) | 907 | 876
  Spit/cough on walls/doors (baseline) | 199 | 257
  Spit/cough on walls/doors (month 6) | 153 | 187

8. Secondary Outcome: Latrine Cleanliness - Cigarette Butts
Description: Assessment by observer in unannounced visit to the shared latrine to determine problems with cleanliness. Observations were made for cigarette butts in toilets. The count of units that had the problem is presented for each problem type.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle. Cubicles that were evaluated were included in the analysis.
Measure: Count of Units; unit: Cubicles
Units Other Than Participants: Cubicles
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Cubicles) | 906 | 916
Cubicles
  Cigarette Butts (baseline) | 95 | 112
  Cigarette Butts (month 6) | 50 | 73

9. Secondary Outcome: Latrine Cleanliness - Waterlogging
Description: Assessment by observer in unannounced visit to the shared latrine to determine problems with cleanliness. Observations were made for waterlogging in toilets. The count of units that had the problem is presented for each problem type.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle. Cubicles that were evaluated were included in the analysis.
Measure: Count of Units; unit: Cubicles
Units Other Than Participants: Cubicles
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Cubicles) | 906 | 916
Cubicles
  Waterlogging (baseline) | 90 | 77
  Waterlogging (month 6) | 35 | 41

10. Secondary Outcome: Latrine Cleanliness - Presence of Household Waste/Waste Wrapped in Polythene
Description: Assessment by observer in unannounced visit to the shared latrine to determine problems with cleanliness. Observations were made for presence of household waste/waste wrapped in polythene. The count of units that had the problem is presented for each problem type.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle. Cubicles that were evaluated were included in the analysis.
Measure: Count of Units; unit: Cubicles
Units Other Than Participants: Cubicles
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Cubicles) | 906 | 916
Cubicles
  Household or polythene-wrapped waste (baseline) | 91 | 43
  Household or polythene-wrapped waste (month 6) | 36 | 26

11. Secondary Outcome: Latrine Cleanliness - Presence of Rags/Sanitary Pads
Description: Assessment by observer in unannounced visit to the shared latrine to determine problems with cleanliness. Observations were made for presence of rags/sanitary pads. The count of units that had the problem is presented for each problem type.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle. Cubicles that were evaluated were included in the analysis.
Measure: Count of Units; unit: Cubicles
Units Other Than Participants: Cubicles
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Cubicles) | 906 | 916
Cubicles
  Rags/Sanitary Pads (baseline) | 43 | 47
  Rags/Sanitary Pads (month 6) | 12 | 23

12. Secondary Outcome: Latrine Cleanliness - Smell of Feces
Description: Assessment by observer in unannounced visit to the shared latrine to determine problems with cleanliness. Observations were made for smell of feces. The count of units that had the problem is presented for each problem type.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle. Cubicles that were evaluated were included in the analysis.
Measure: Count of Units; unit: Cubicles
Units Other Than Participants: Cubicles
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Cubicles) | 906 | 916
Cubicles
  Smell of Feces (baseline) | 521 | 504
  Smell of Feces (month 6) | 319 | 382

13. Secondary Outcome: Latrine Cleanliness - Smell of Urine
Description: Assessment by observer in unannounced visit to the shared latrine to determine problems with cleanliness. Observations were made for smell of urine. The count of units that had the problem is presented for each problem type.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle. Cubicles that were evaluated were included in the analysis.
Measure: Count of Units; unit: Cubicles
Units Other Than Participants: Cubicles
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Cubicles) | 906 | 916
Cubicles
  Smell of Urine (baseline) | 463 | 516
  Smell of Urine (month 6) | 264 | 333

14. Secondary Outcome: Latrine Cleanliness - Smell of Cigarettes
Description: Assessment by observer in unannounced visit to the shared latrine to determine problems with cleanliness. Observations were made for smell of cigarettes. The count of units that had the problem is presented for each problem type.
Time Frame: Assessed at 6 months post intervention
Population: Shared latrines may have had more than one cubicle. Cubicles that were evaluated were included in the analysis.
Measure: Count of Units; unit: Cubicles
Units Other Than Participants: Cubicles
Arm/Group | Behavior Change | Control Arm
Number analyzed (Participants) | 609 | 605
Number analyzed (Cubicles) | 906 | 916
Cubicles
  Smell of cigarettes (baseline) | 83 | 111
  Smell of cigarettes (month 6) | 54 | 65

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Behavior Change | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/609 | 0/605
Serious Adverse Events (participants affected / at risk) | 0/609 | 0/605
Other Adverse Events (participants affected / at risk) | 0/609 | 0/605

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No